CLINICAL TRIAL: NCT06967129
Title: Evaluation of Daily Disposable Toric Soft Lenses Manufactured With an Alternative Hydration Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6590
Record Dates: First submitted 2025-04-22; First posted 2025-05-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test/Control (Experimental): Eligible subjects will be randomized to the Test/Control sequence, to wear the Test Lens followed by the Control Lens bilaterally for approximately 1-week each in a daily disposable modality with a washout period of approximately 1-week between wear periods.
  Interventions: Device: Investigational daily disposable, soft, toric lenses manufactured on 4th Generation Technology (4GT) lines with extended mini-stack hydration using propylene glycol (PG) as the hydration solvent.; Device: ACUVUE® Oasys 1-Day for Astigmatism (AO1DfA) soft contact lenses manufactured on 3rd Generation Technology (3GT) legacy lines using isopropyl alcohol (IPA) as the hydration solvent.
- Control/Test (Experimental): Eligible subjects will be randomized to the Control/Test sequence, to wear the Control Lens followed by the Test Lens bilaterally for approximately 1-week each in a daily disposable modality with a washout period of approximately 1-week between wear periods.
  Interventions: Device: Investigational daily disposable, soft, toric lenses manufactured on 4th Generation Technology (4GT) lines with extended mini-stack hydration using propylene glycol (PG) as the hydration solvent.; Device: ACUVUE® Oasys 1-Day for Astigmatism (AO1DfA) soft contact lenses manufactured on 3rd Generation Technology (3GT) legacy lines using isopropyl alcohol (IPA) as the hydration solvent.

INTERVENTIONS:
Device: Investigational daily disposable, soft, toric lenses manufactured on 4th Generation Technology (4GT) lines with extended mini-stack hydration using propylene glycol (PG) as the hydration solvent. — Test Lens
Device: ACUVUE® Oasys 1-Day for Astigmatism (AO1DfA) soft contact lenses manufactured on 3rd Generation Technology (3GT) legacy lines using isopropyl alcohol (IPA) as the hydration solvent. — Control Lens

SUMMARY:
This is a prospective, multi-site, dispensing, randomized, controlled, double-masked, bilateral wear, 2x2 crossover study to evaluate the safety and effectiveness of the test lens.

ELIGIBILITY:
Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 2 days per week during last 30 days.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. In both eyes, have astigmatic refractive error suitable for correction with the toric contact lens powers available in this study:

   1. Sphere powers (DS) -1.50 through -4.00 (inclusive) in 0.25 steps
   2. Cylinder powers (DC) -0.75 and -1.25
   3. Axes (°) 170, 180, 10, 80, 90, 100
7. Have best corrected monocular distance visual acuity of 20/30 or better in each eye.

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have an ocular infection of any type.
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
6. Be currently wearing monovision or multifocal contact lenses.
7. Be currently wearing lenses in an extended wear modality.
8. Have a history of strabismus or amblyopia.
9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, Photorefractive Keratectomy [PRK], Laser-Assisted in Situ Keratomileusis [LASIK], iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 281 (Actual)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Distance (4m) Monocular High Luminance High Contrast (HLHC) logMAR Visual Acuity (VA) | At each 1-week follow-up per wear period
  VA will be assessed monocularly under HLHC conditions at a test distance of 4 meters using ETDRS Charts.
Toric Lens Orientation | At baseline per wear period
  Toric lens orientation (scribe mark position relative to 6 o'clock) will be assessed for each eye at 15 minutes after lens insertion. Toric lens orientation will be used to define a binary endpoint, i.e. the percentage of eyes that achieve absolute toric lens rotation ≤ 10°.
Lens Rotational Stability with Blinks | At baseline per wear period
  Rotational stability will be assessed for each eye at least 15 minutes after lens insertion. Lens rotational stability with blinks will be defined as a binary endpoint, the percentage of eyes that achieve rotational stability with blinks ≤ 5°.
Percentage of eyes with Grade 3 or higher SLFs relating to the test lens | Up to 3-week follow-up
  SLFs (Grade 3 or higher) related to study lens wear for the test lens will be assessed for each eye at all study visits (scheduled and unscheduled). SLFs will be evaluated and graded using the FDA Grading scale from 0 to 4, where Grade 0 represents the absence of findings and 1 to 4 representing successively worse findings. The percentage of eyes with Grade 3 or higher SLF will be analyzed and will include corneal infiltrates.
Percentage of eyes with acceptable lens fitting while wearing the test lens | Up to 3-week follow-up
  Acceptable lens fit will be assessed at all study visits (scheduled and unscheduled) for each subject eye and used to define a binary endpoint, i.e. the percentage of eyes that achieve acceptable lens fit while wearing the test lens.
  Lens fit will be deemed unacceptable if any one of the following criteria are met:
  * limbal exposure at primary gaze or with extreme eye movement.
  * edge lift.
  * excessive movement on blink in primary gaze.
  * insufficient movement in all three of the following conditions: primary gaze, up gaze, and push up test.

SECONDARY OUTCOMES:
Subjective Overall Comfort | At each 1-week follow-up per wear period
  Subjective overall Comfort scores will be assessed using the CLUE questionnaire. CLUE™ is a validated, patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, for wearers between 18 to 65 years of age. CLUE™ scores are derived using Item Response Theory (IRT) and follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Subjective Overall Quality of Vision | At each 1-week follow-up per wear period
  Subjective Overall Quality of Vision scores will be assessed using the CLUE questionnaire. CLUE™ is a validated, patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, for wearers between 18 to 65 years of age. CLUE™ scores are derived using Item Response Theory (IRT) and follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Subjective Overall Handling | At each 1-week follow-up per wear period
  Subjective Overall Handling scores will be assessed using the CLUE questionnaire. CLUE™ is a validated, patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, for wearers between 18 to 65 years of age. CLUE™ scores are derived using Item Response Theory (IRT) and follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (20):
- United States (20):
  - James R. Dugue, Optometrist, Mission Viejo, California
  - Scripps Poway Eyecare & Optometry, San Diego, California
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Pearson Research Center PA, Longwood, Florida
  - Maitland Vision Centers - North Orlando Ave, Maitland, Florida
  - Mid-State Eye, Clinton, Illinois
  - Franklin Park Eye Center, P.C., Franklin Park, Illinois
  - Kannarr Eye Care - 101 North Broadway, Pittsburg, Kansas
  - Complete Eye Care of Medina, Medina, Minnesota
  - Advanced Eyecare - Raytown, MO, Raytown, Missouri
  - The Koetting Associates, St Louis, Missouri
  - ABQ Eye Care, Albuquerque, New Mexico
  - Spectrum Eye Care, Jamestown, New York
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - Professional Vision Care Inc. - Westerville, Westerville, Ohio
  - Optometry Group, PLLC, Memphis, Tennessee
  - Total Eye Care, Memphis, Tennessee
  - Tyler Eye Associates, Tyler, Texas
  - Clarke EyeCare Center, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu